CLINICAL TRIAL: NCT04252521
Title: Intravenous Metoclopramide Versus Dexketoprofen Trometamol Versus Metoclopramide+ Dexketoprofen Trometamol in Acute Migraine Attack in the Emergency Department: a Randomized Double-blind Controlled Trial
Brief Title: Intravenous Metoclopramide Versus Dexketoprofen Trometamol Versus Metoclopramide+ Dexketoprofen Trometamol in Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Umut Gulacti, Clinical Associate Professor, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 66175679-514.04.01
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Metoclopramide; dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- metoclopramide+ dexketoprofen trometamol (Active Comparator): 10 mg metoclopramide+ 50 mg dexketoprofen trometamol
  Interventions: Drug: metoclopramide+dexketoprofen trometamol
- metoclopramide (Experimental): 10 mg metoclopramide
  Interventions: Drug: metoclopramide
- dexketoprofen trometamol (Experimental): 50 mg dexketoprofen trometamol
  Interventions: Drug: dexketoprofen trometamol

INTERVENTIONS:
Drug: metoclopramide — 10 mg Metpamid in 100 ml normal saline solution
  Other Names: Metpamid (metoclopramide)
  Arms: metoclopramide
Drug: dexketoprofen trometamol — 50 mg dexketoprofen trometamol in 100 ml normal saline solution
  Other Names: Metadem (dexketoprofen trometamol)
  Arms: dexketoprofen trometamol
Drug: metoclopramide+dexketoprofen trometamol — 10 mg metoclopramide+50 mg dexketoprofen trometamol in 100 ml normal saline solution
  Other Names: Metpamid+Metadem
  Arms: metoclopramide+ dexketoprofen trometamol

SUMMARY:
Acute headache is one of the most common reasons for presentation to the emergency department (ED), accounting for 2-3% of all emergency visits. Migraine is a disorder of the central nervous system characterized by a moderate or severe headache, which is generally associated with nausea and/or sensitivity to light and sound, interfering with daily activities.

DETAILED DESCRIPTION:
Study objective: The objective of this study is to determine the analgesic efficacy and safety of intravenous, single-dose metoclopramide versus dexketoprofen trometamol versus metoclopramide+ dexketoprofen trometamol in patients presenting with acute migraine attack to the emergency department (ED).

Methods of Measurements:

This single-center, randomized, double-blind study will be conducted in a tertiary care ED. Eligible patients who met the migraine criteria of the International Headache Society will be randomized to receive 10 mg intravenous metoclopramide, 50 mg intravenous dexketoprofen trometamol, or 50 mg dexketoprofen trometamol + 10 mg metoclopramide.

Subjects reported pain intensity on both a 100-mm visual analogue scale (VAS) (limited by 'no pain' and 'the worst pain') will be used for pain measurement at baseline, after 15 and 30 min. The primary outcome measure is the changes in the VAS scores at the 15th and 30th minutes of treatment. The secondary outcome measures are the presence of adverse effects and the requirement of rescue medicine.

Primary Data Analysis:

The study was planned as a superiority trial. The difference in the VAS values between the groups was assumed to detect 21.4 mm and the standard deviation (SD) value as 2.8 mm, and thus the minimum required the number of patients for each group was calculated as 27 at the alpha-critical value of 0.05 and power of 80%. All the analyses were implemented according to the intention to treat analysis. Differences between time intervals within groups and between groups and statistical significance were expressed by 95% confidence intervals (95% CI).

ELIGIBILITY:
Inclusion Criteria:

-Patients aged 18 and over with acute headache who met the diagnostic criteria of the International Headache Association (9) for the diagnosis of migraine

Exclusion Criteria:

* Patients who refused to participate in the study
* Patients that took any analgesic medication within six hours before presentation to ED Patients with any additional organic pathology (e.g., hypertension, hypoglycemia, chronic kidney failure, and intracranial masses) pregnant women hemodynamically unstable patients patients with an allergy to the drugs used in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Change of the intensity of pain | 15 minutes and 30 minutes after the study drug administered
  Pain intense will be measured by 100 mm visual analog scale (Zero; no pain and 100 mm; the worst pain) after 15th and 30th minutes later after the study drug administered

SECONDARY OUTCOMES:
Adverse events | 30 minutes after
  30 minutes after the study drug administered
need to rescue medication | 30 minutes after
  30 minutes after the study drug administered

CONTACTS AND LOCATIONS:
Overall Officials: Umut Gülaçtı, Principal Investigator — Adiyaman University of Medical Faculty
Locations (1):
- Adiyaman University Research Hospital, Adıyaman, Central, Turkey (Türkiye)

REFERENCES:
- [Background] Egerton-Warburton D, Meek R, Mee MJ, Braitberg G. Antiemetic use for nausea and vomiting in adult emergency department patients: randomized controlled trial comparing ondansetron, metoclopramide, and placebo. Ann Emerg Med. 2014 Nov;64(5):526-532.e1. doi: 10.1016/j.annemergmed.2014.03.017. Epub 2014 May 10. PMID 24818542
- [Background] Yang B, Xu Z, Chen L, Chen X, Xie Y. The efficacy of dexketoprofen for migraine attack: A meta-analysis of randomized controlled studies. Medicine (Baltimore). 2019 Nov;98(46):e17734. doi: 10.1097/MD.0000000000017734. PMID 31725614
- [Derived] Yavuz E, Gulacti U, Lok U, Turgut K. Intravenous metoclopramide versus dexketoprofen trometamol versus metoclopramide+ dexketoprofen trometamol in acute migraine attack in the emergency department: A randomized double-blind controlled trial. Am J Emerg Med. 2020 Nov;38(11):2254-2258. doi: 10.1016/j.ajem.2020.04.038. Epub 2020 Apr 15. PMID 32359776